CLINICAL TRIAL: NCT05492474
Title: Cranial Ultrasound for Prehospital ICH Diagnosis (CUPID_EMS)
Brief Title: Cranial Ultrasound for Prehospital ICH Diagnosis
Acronym: CUPID_EMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB00077652
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Intracerebral Hemorrhage; Acute Ischemic Stroke
Keywords: computed tomography (CT) scan
MeSH Terms: conditions — Cerebral Hemorrhage; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Any patient deemed to have a stroke like presentation or possibility of brain hemorrhage in the clinical judgement of the EMS provider and a decision to transfer the patient to the nearest ED for further evaluation has been made
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cranial Point of Care Ultrasound (Experimental): Cranial ultrasound involves 2-dimensional B mode imaging of the brain parenchyma in the axial plane
  Interventions: Procedure: Cranial Point of Care Ultrasound

INTERVENTIONS:
Procedure: Cranial Point of Care Ultrasound — Cranial ultrasound involves 2-dimensional B mode imaging of the brain parenchyma in the axial plane using a 1-2 MHz probe through the thin temporal bone. Upload of cPOCUS images will occur over DICOM® based Health Insurance Portability and Accountability Act (HIPAA) compliant platforms accessible via Cloud. Currently all handheld machines use Tricefy® or their own cloud based remote image access application.

SUMMARY:
To evaluate the feasibility of Emergency Medical System (EMS)-performed cPOCUS in the field for diagnosis of acute Intracerebral hemorrhage (ICH)

DETAILED DESCRIPTION:
With the over-arching goal of achieving early diagnosis of Intracerebral hemorrhage (ICH) with cPOCUS, this study hypothesizes that (a) Emergency Medical System (EMS) personnel can competently perform cPOCUS in the field in a timely fashion in a large majority of stroke patients; (b) acquired POCUS images can be successfully and securely transmitted for a remote physician interpretation in a timely manner; and (c) cPOCUS will have a greater sensitivity and specificity than clinical scores as a screening tool for ICH identification in pre-hospital settings.

ELIGIBILITY:
Inclusion Criteria:

* Any patient deemed to have a stroke like presentation or possibility of brain hemorrhage in the clinical judgement of the Emergency Medical Services (EMS) provider and a decision to transfer the patient to the nearest Emergency Department (ED) for further evaluation has been made will be eligible for the study
* 18 years old or older
* transfer initiated by EMS to the ED for further evaluation
* performing ultrasound will not interfere with the care or triage as part of routine care

Exclusion Criteria:

* less than 18 years old
* incarcerate patients
* penetrating cranial/head trauma or scalp wound
* any patient where performing ultrasound will interfere with the care
* patients who decide not to be transported to ED

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Success Rate for cPOCUS Exams | Year 1
  cPOCUS will be attempted and performed on about 1000 patients over 12 months by 30 EMS providers

CONTACTS AND LOCATIONS:
Overall Officials: Aarti Sarwal, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal

DOCUMENTS (1):
  • Informed Consent Form (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT05492474/ICF_000.pdf